CLINICAL TRIAL: NCT03322683
Title: Vacuum Myofascial Therapy Device for Non-specific Neck Pain. A Single Blind Randomized Clinical Trial
Brief Title: Treatment of Cervical Syndrome With Physium Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: physium therapy
Record Dates: First submitted 2017-10-18; First posted 2017-10-26 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Cervical Syndrome
Keywords: Neck Pain; Physical Therapy Modalities; Massage; Manual Therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CLINICAL TRIAL WITH BLIND EVALUATION BY THIRD PARTIES, LONGITUDINAL AND PROSPECTIVE.
Who Masked: Investigator
Masking Description: Blind researcher
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): The intervention for this group consisted of 5 massage sessions with the PHYSIUM device for a month.
  Interventions: Procedure: Physiotherapy treatment with physium device.
- CONTROL GROUP (Experimental): The multimodal physical therapy program includes 10 sessions of:
  * ultrasound pulsatil therapy (US) for 10 minutes.
  * transcutaneous electric nerve stimulation (TENS) for 20 minutes.
  * massage for 20 minutes.
  Interventions: Procedure: Conventional physiotherapy treatmen

INTERVENTIONS:
Procedure: Physiotherapy treatment with physium device. — This group will treated five times with the analgesic program of physium therapy. Each maneuver was performed once per session by slow and progressive. The whole procedure lasted no more than 45 minutes.
  Arms: EXPERIMENTAL GROUP
Procedure: Conventional physiotherapy treatmen — The PT group will treated during two weeks (ten days/week) with ultrasound therapy (US), transcutaneous electric nerve stimulation (TENS) and massage, in this order. Ultrasound will applied in pulse mode at an intensity of 1 megahertz for 10 minutes in the sub-occipital region and the vicinity of the trapezius muscles. TENS will applied with a pulse duration of 250 microseconds at a frequency of 80 Hertz for 20 minutes in the sub-occipital region and the trapezoids. Deep massage was applied at a slow speed for 20 minutes using sliding neutral creams. Massage therapy included gliding and kneading techniques applied over trapezius (upper, lower and middle fibers), splenius capitis and levator scapulae muscles with a therapeutic intention.
  Arms: CONTROL GROUP

SUMMARY:
This study aim to investigate the effects of physium therapy for improving pressure pain thresholds (PPTs), range of motion,Neck Disability Index, the multidimensional health related quality of life (SF-12) and the multidimensional health related quality of life and pain in patients with mechanical neck pain (NP).

DETAILED DESCRIPTION:
Fifty-four participants with NP will randomly allocated to either an physium therapy (five sessions) or a physical therapy (PT) groups (ten sessions) during two weeks. Multimodal PT program included: ultrasound therapy (US), transcutaneous electric nerve stimulation (TENS) and massage. Visual Analogue Scale (VAS), Neck Disability Index ( NDI), range of motion and (CROM), Questionnaire SF-12 and PPTs in sub-occipital and upper trapezius muscles were measured at baseline, at the end of treatment and at 1 month follow-up. T-tests and a repeated-measures multivariate analysis of variance (RM-MANOVA) were used for VAS, CROM and PPTs, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes,
* Aged between 20 and 60 years, in an
* Active state of pain and diagnosed with a month of evolution.

Exclusion Criteria:

- Patients who are pregnant, have pacemaker and those Surgically operated cervical spine - - Patients who have been treated with myofascial therapy a month earlier.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
The intensity of cervical pain | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.

SECONDARY OUTCOMES:
The intensity of cervical pain | Four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.
Active cervical range of motion | Baseline and four weeks.
  Measured by goniometer type crom
Pressure pain thresholds in cervical trigger points | Baseline and four weeks
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline, Pain TestTM, Wagner Instruments). The clinimetric properties of this instrument have been evaluated previously. The PPT will the point at which pressure elicited pain and will presented as kilograms per square centimeter. All measurements will be conducted by the same well-trained physician.
The multidimensional health related quality of life | Baseline and four weeks
  Questionnaire SF 12
This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. | Baseline and four weeks.
  Neck Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodriguez Huguet, Principal Investigator — University of Cadiz
Locations (1):
- Clínica Pastoriza, El Puerto de Santa María, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Leaver AM, Maher CG, McAuley JH, Jull G, Latimer J, Refshauge KM. People seeking treatment for a new episode of neck pain typically have rapid improvement in symptoms: an observational study. J Physiother. 2013 Mar;59(1):31-7. doi: 10.1016/S1836-9553(13)70144-9. PMID 23419913
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Palmlof L, Skillgate E, Alfredsson L, Vingard E, Magnusson C, Lundberg M, Holm LW. Does income matter for troublesome neck pain? A population-based study on risk and prognosis. J Epidemiol Community Health. 2012 Nov;66(11):1063-70. doi: 10.1136/jech-2011-200783. Epub 2012 Mar 12. PMID 22412154
- [Background] Noormohammadpour P, Mansournia MA, Koohpayehzadeh J, Asgari F, Rostami M, Rafei A, Kordi R. Prevalence of Chronic Neck Pain, Low Back Pain, and Knee Pain and Their Related Factors in Community-Dwelling Adults in Iran: A Population-based National Study. Clin J Pain. 2017 Feb;33(2):181-187. doi: 10.1097/AJP.0000000000000396. PMID 27258995
- [Background] De Pauw R, Coppieters I, Kregel J, De Meulemeester K, Danneels L, Cagnie B. Does muscle morphology change in chronic neck pain patients? - A systematic review. Man Ther. 2016 Apr;22:42-9. doi: 10.1016/j.math.2015.11.006. Epub 2015 Dec 11. PMID 26724855
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Cook AJ, Wellman RD, Cherkin DC, Kahn JR, Sherman KJ. Randomized clinical trial assessing whether additional massage treatments for chronic neck pain improve 12- and 26-week outcomes. Spine J. 2015 Oct 1;15(10):2206-15. doi: 10.1016/j.spinee.2015.06.049. Epub 2015 Jun 19. PMID 26096474
- [Background] Liptan G, Mist S, Wright C, Arzt A, Jones KD. A pilot study of myofascial release therapy compared to Swedish massage in fibromyalgia. J Bodyw Mov Ther. 2013 Jul;17(3):365-70. doi: 10.1016/j.jbmt.2012.11.010. Epub 2013 Jan 3. PMID 23768283
- [Background] Yuan SL, Matsutani LA, Marques AP. Effectiveness of different styles of massage therapy in fibromyalgia: a systematic review and meta-analysis. Man Ther. 2015 Apr;20(2):257-64. doi: 10.1016/j.math.2014.09.003. Epub 2014 Oct 5. PMID 25457196
- [Background] Serrano-Aguilar P, Kovacs FM, Cabrera-Hernandez JM, Ramos-Goni JM, Garcia-Perez L. Avoidable costs of physical treatments for chronic back, neck and shoulder pain within the Spanish National Health Service: a cross-sectional study. BMC Musculoskelet Disord. 2011 Dec 21;12:287. doi: 10.1186/1471-2474-12-287. PMID 22188790
- [Background] Cagnie B, Castelein B, Pollie F, Steelant L, Verhoeyen H, Cools A. Evidence for the Use of Ischemic Compression and Dry Needling in the Management of Trigger Points of the Upper Trapezius in Patients with Neck Pain: A Systematic Review. Am J Phys Med Rehabil. 2015 Jul;94(7):573-83. doi: 10.1097/PHM.0000000000000266. PMID 25768071
- [Background] Bervoets DC, Luijsterburg PA, Alessie JJ, Buijs MJ, Verhagen AP. Massage therapy has short-term benefits for people with common musculoskeletal disorders compared to no treatment: a systematic review. J Physiother. 2015 Jul;61(3):106-16. doi: 10.1016/j.jphys.2015.05.018. Epub 2015 Jun 17. PMID 26093806
- [Background] Fletcher JP, Bandy WD. Intrarater reliability of CROM measurement of cervical spine active range of motion in persons with and without neck pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):640-5. doi: 10.2519/jospt.2008.2680. PMID 18827326
- [Background] Lopez-Lopez A, Alonso Perez JL, Gonzalez Gutierez JL, La Touche R, Lerma Lara S, Izquierdo H, Fernandez-Carnero J. Mobilization versus manipulations versus sustain apophyseal natural glide techniques and interaction with psychological factors for patients with chronic neck pain: randomized controlled trial. Eur J Phys Rehabil Med. 2015 Apr;51(2):121-32. Epub 2014 Oct 9. PMID 25296741
- [Background] Bonilla D, Hortalá G, Temporal D, Carré Llopis C. PHYSIUM in the treatment of pain in patients with chronic low back pain. FisioGlía. 2015;2(3):50-55.
- [Background] Canadell G. Effectiveness of PHYSIUM Massage in chronic neck pain in patients not responding to the standard physiotherapy. MC Health & Medical Publishing. 2011;1.